CLINICAL TRIAL: NCT03456947
Title: Research of Pregabalin Stabilize Cardiovascular Response to Laryngoscopy and Tracheal Intubation of Patients Under General Anesthesia
Brief Title: Pregabalin Stabilize Cardiovascular Response to Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWW-PRBL-2017
Record Dates: First submitted 2018-02-27; First posted 2018-03-07 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Effect of Laryngoscopy and Tracheal Intubation
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (No Intervention): the patients receive routine preoperative preparation without having Pregabalin
- Pregabalin150mg group (Experimental): the patients receive 150mg pregabalin 60 minutes prior to the surgery
  Interventions: Drug: Pregabalin
- Pregabalin300mg group (Experimental): the patients receive 300mg pregabalin 60 minutes prior to the surgery
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — the patients receive 150mg or 300mg pregabalin 60 minutes prior to the surgery
  Arms: Pregabalin150mg group; Pregabalin300mg group

SUMMARY:
The purpose of the study is to evaluate whether Pregabalin is safe and effective in stabilizing cardiovascular response to laryngoscopy and tracheal intubation of patients under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists(ASA) grade I and II scheduled for elective surgery

Exclusion Criteria:

* patient refusal.
* patients with serious chronic kidney, liver, lungs, or cardiovascular diseases.
* allergy to any of the study medications.
* patients taking sedation or antihypertensive medications.
* suspected difficult intubation or intubation time more than 22s.
* pregnant or breastfeeding women.
* BMI>30.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
heart rate | heart rate 3 minutes after intubation
  effect of 300mg pregabalin, 150mg pregabalin premedication versus control group on the heart rate due to laryngoscopy and tracheal intubation

SECONDARY OUTCOMES:
Mean arterial blood pressure | baseline mean arterial blood pressure before drug administration, heart rate before intubation, heart rate after 0 minute, 1minute, 3minutes, 5 minutes, 7minutes, 10minutes after intubation and before skin incision
  effect of 300mg pregabalin, 150mg pregabalin premedication versus control group on the Mean arterial blood pressure due to laryngoscopy and tracheal intubation
systolic blood pressure | baseline systolic blood pressure before drug administration, heart rate before intubation, heart rate after 0 minute, 1minute, 3minutes, 5 minutes, 7minutes, 10minutes after intubation and before skin incision
  effect of 300mg pregabalin, 150mg pregabalin premedication versus control group on the systolic blood pressure due to laryngoscopy and tracheal intubation
diastolic blood pressure | baseline diastolic blood pressure before drug administration, heart rate before intubation, heart rate after 0 minute, 1minute, 3minutes, 5 minutes, 7minutes, 10minutes after intubation and before skin incision
  effect of 300mg pregabalin, 150mg pregabalin premedication versus control group on the diastolic blood pressure due to laryngoscopy and tracheal intubation
Ramsay score | baseline Ramsay score before drug administration and Ramsay score before intubation
  Ramsay score of 300mg pregabalin, 150mg pregabalin premedication versus
Incidence of all clinical adverse events | 1hour after surgery
  The occurrence of dizziness, nausea, vomit and allergy

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Principal Investigator — Zhongshan Hospital Qinpu Branch, Fudan University, Shanghai

REFERENCES:
- [Derived] Chen W, Huang H, Yang C, Hu X, Bao F, Jiang H. Preoperative Low-dose and High-dose Pregabalin and Cardiovascular Response to Endotracheal Intubation: A Prospective, Randomized, Single-blind, Controlled Study in China. Clin Ther. 2019 Jan;41(1):68-77. doi: 10.1016/j.clinthera.2018.11.006. Epub 2018 Dec 13. PMID 30553555